CLINICAL TRIAL: NCT05927558
Title: Salvage Treatment With Glofitamab in Patients Affected by Relapsed/Refractory Non-Hodgkin B-cell Lymphoma: a GIMEMA-FIL Study
Brief Title: Salvage Treatment With Glofitamab in R/R B-NHL: a GIMEMA-FIL Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: IMM0123
Record Dates: First submitted 2023-06-22; First posted 2023-07-03 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: B-cell Non Hodgkin Lymphoma; Relapse; Refractory Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Recurrence; Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to evaluate the anti-lymphoma activity of glofitamab, administered according to the Compassionate Use Program, in relapsed/refractory B-NHL patients. The main question it aims to answer is the rate of patients in complete response.

DETAILED DESCRIPTION:
This is an observational multicenter study aimed at assessing the anti-lymphoma activity of glofitamab in relapsed/refractory B cell non-Hodgikin lymphoma patients treated according to the Compassionate Use Program in Italy between March 2022 and September 2023. Patients will be observed for a minimum of 12 months after the last glofitamab administration.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who received glofitamab according to Compassionate Use Program AG42296
2. Age > 18 years
3. Patients who received at least one dose of glofitamab between March 2022 and September 2023 in the context of the compassionate use program and who completed at least 1 year of observation after last glofitamab administration unless the patient died or was lost to follow up
4. Patients who provided their consent according to local regulation to collect their data for study purposes, dead patients or patients lost to follow up for which any attempt has been made to collect their consent, according to local regulation on data privacy

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with refractory/relapsed B-cell non-Hodgkin lymphoma treated in Italy according to the Compassionate Use Program between March 2022 and September 2023
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2023-12-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Rate of patients in complete response | 6 months
  Effectiveness of glofitamab in terms of complete response

CONTACTS AND LOCATIONS:
Locations (1):
- Ematologia Istituto Nazionale Tumori, Milan, Italy